CLINICAL TRIAL: NCT00289835
Title: Sealing Moderate Coronary Saphenous VEin Graft LEsions With the Paclitaxel-eluting Stent (Taxus) as a New Approach to Maintain Vein Graft Patency and Reduce Cardiac Events: a Pilot Intravascular Ultrasound Study.
Brief Title: Treatment of Moderate Vein Graft Lesions With Paclitaxel Drug Eluting Stents: The VELETI Trial
Acronym: VELETI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Laval University (Other)
Collaborators: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Laval-VG-01
Record Dates: First submitted 2006-02-09; First posted 2006-02-10 (Estimated); Last update posted 2011-11-24 (Estimated); Status verified 2008-10

CONDITIONS: Coronary Artery Bypass Grafting
Keywords: Coronary Artery Bypass Grafting; Drug Eluting Stent; Saphenous Vein Graft

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- PCI-stenting (Experimental): Stenting the moderate SVG lesion with the paclitaxel stent
  Interventions: Device: Paclitaxel eluting stent
- Standard medical treatment (Other)
  Interventions: Device: Paclitaxel eluting stent

INTERVENTIONS:
Device: Paclitaxel eluting stent — Patients are randomized to either stenting the moderate SVG lesion with the paclitaxel stent or standard medical treatment
  Other Names: Taxus (paclitaxel eluting stent)

SUMMARY:
HYPOTHESIS

1. Sealing moderate SVG lesions with the TAXUS stent prevents SVG atherosclerosis progression as evaluated by IVUS.
2. Sealing moderate SVG lesions with the TAXUS stent does not accelerate SVG atherosclerosis in the angiographically non-diseased segments of the SVG as evaluated by IVUS.

OBJECTIVES

1. To determine the effect of stenting moderate SVG lesions with the paclitaxel-eluting stent in comparison with medical treatment on limiting SVG disease progression as evaluated by IVUS.
2. To evaluate by IVUS the effect of stenting moderate SVG lesions with the paclitaxel-eluting stent in comparison with medical treatment on atherosclerosis progression in angiographically non-diseased SVGs segments.

DETAILED DESCRIPTION:
This will be a prospective randomized study assessing the efficacy of stenting moderate SVG lesions with the taxus stent in the prevention of atherosclerosis progression of SVGs as evaluated by IVUS. Patients with previous coronary bypass surgery with SVG implantation undergoing coronary angiography by clinical indication will be screened. If the patient has a moderate lesion at any level of the SVGs it will be includable in the study. After inclusion, the patients will be randomized to either stenting the moderate SVG lesion with the taxus stent or standard medical treatment. The use of a filter wire during dilation will be strongly recommended. Following this procedure, all patients will have clinical controls at 1 month and at 6 months and an angiographic and IVUS control study at 1 year follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Written and signed informed consent.
* Patients ≥18 years old.
* Clinical indication for cardiac catheterization and SVG angiography.
* Presence of at least one SVG lesion of 30% to 70% diameter stenosis by visual estimation which is (are) not the culprit lesion (s) responsible for the clinical syndrome of the patient.

Exclusion Criteria:

* Ejection fraction <20%.
* Renal insufficiency with creatinine > 250 mg/dl.
* Presence of more than 3 moderate SVG stenosis or significant diffuse SVG disease.
* Unsuccessful angioplasty (residual stenosis >30% and/or TIMI flow <3) of any other lesion treated during the same procedure.
* Coronary angioplasty of the target SVG in the past.
* Cardiogenic shock .
* Remaining lesion (s) with a treatment planned within the following year.
* Pregnancy.
* Contraindication to aspirin and/or clopidogrel treatment.
* Allergy to paclitaxel.
* Any disease with a limiting life-expectancy (to less than 2 years).
* Definite presence or high suspicion of thrombus or ulceration in the target lesion.
* Target lesion located in the same SVG than the culprit lesion (if present) and the distance between the target lesion and the most proximal or distal part of the stent implanted at the culprit lesion is < 4 cm.
* Vein graft diameter < 2.5 mm.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2006-02; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Ultrasound lumen area and minimal lumen diameter at follow-up at the tomographic section showing the most severe stenosis, comparing stented vs medically treated SVGs lesions | 12 months
Change between baseline and follow-up in ultrasound lumen area and minimal lumen diameter (% and absolute value) at the tomographic section showing the most severe stenosis, comparing stented vs medically treated SVGs lesions | 12 months
Change in atheroma volume (% and absolute value) as evaluated by IVUS between baseline and follow-up in an angiographically non-diseased 40 mm segment (excluding the target lesion), comparing stented vs medically treated SVGs | 12 months

SECONDARY OUTCOMES:
Cumulative incidence of clinical events (cardiovascular death, myocardial infarction, repeat revascularization) at 12 months follow-up | 12 months
SVG occlusion rate, lesion/stent late loss, minimal lumen diameter, and % diameter stenosis as assessed by angiography at 12 months follow-up | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Josep Rodes-Cabau, MD, Principal Investigator — Laval Hospital Research Center; Olivier F Bertrand, MD, PhD, Principal Investigator — Laval Hospital Research Center; Robert Delarocheliere, MD, Principal Investigator — Laval Hospital Research Center
Locations (1):
- Laval Hospital, Québec, Quebec, Canada

REFERENCES:
- [Derived] Rodes-Cabau J, Bertrand OF, Larose E, Dery JP, Rinfret S, Urena M, Jerez M, Nombela-Franco L, Ribeiro HB, Allende R, Proulx G, Nguyen CM, Boudreault JR, Rouleau J, Roy L, Gleeton O, Barbeau G, Noel B, Cote M, Despres JP, Dagenais GR, DeLarochelliere R. Five-year follow-up of the plaque sealing with paclitaxel-eluting stents vs medical therapy for the treatment of intermediate nonobstructive saphenous vein graft lesions (VELETI) trial. Can J Cardiol. 2014 Jan;30(1):138-45. doi: 10.1016/j.cjca.2013.11.002. Epub 2013 Nov 6. PMID 24365196
- [Derived] Rodes-Cabau J, Bertrand OF, Larose E, Dery JP, Rinfret S, Bagur R, Proulx G, Nguyen CM, Cote M, Landcop MC, Boudreault JR, Rouleau J, Roy L, Gleeton O, Barbeau G, Noel B, Courtis J, Dagenais GR, Despres JP, DeLarochelliere R. Comparison of plaque sealing with paclitaxel-eluting stents versus medical therapy for the treatment of moderate nonsignificant saphenous vein graft lesions: the moderate vein graft lesion stenting with the taxus stent and intravascular ultrasound (VELETI) pilot trial. Circulation. 2009 Nov 17;120(20):1978-86. doi: 10.1161/CIRCULATIONAHA.109.874057. Epub 2009 Nov 2. PMID 19884468